CLINICAL TRIAL: NCT06919770
Title: Use of a Taurolidine Containing Antimicrobial Wash to Reduce Prosthetic Device Infection After Trauma Surgery
Acronym: Prosafeti
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hendrik Bonnemeier, coordinating Principal investigator, University of Kiel
Other Study IDs: CUX-1
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Osteosynthesis; Infection Prevention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A taurolidine-based antimicrobial solution, was evaluated for its safety and efficacy in preventing infections associated with prosthetic materials, such as joint replacements, plates, nails, and screws. This prospective observational study compared Taurolidine to infection rates from scientific literature.

DETAILED DESCRIPTION:
During any invasive procedure involving prosthetic materials at the corresponding author's institution, the surgical site was irrigated, and all accessible hardware (including nails, screws, plates, and prosthetic joint replacement therapy devices) was wiped with Taurolidine. Only procedures performed between 01/01/2022 and 01/10/2023, where Taurolidine was applied, were included in the analysis.

Patients who underwent multiple procedures were censored for the last treatment group and reassigned at the next procedure. Preoperative antibiotic prophylaxis was administered according to institutional guidelines, and no additional intraoperative antimicrobial agents were used aside from Taurolidine.

The primary endpoint was the occurrence of a major infection within three months post-procedure, defined as:

1. Infection necessitating revision procedure,
2. A requirement for prolonged antibiotic therapy, or
3. Infection leading to mortality. Secondary endpoints included infections beyond three months, adverse events potentially related to the antimicrobial solution, procedural complications (i.e., hematoma formation, nerval lesions, etc), and mortality during all follow-up.

ELIGIBILITY:
Inclusion Criteria:

* requires osteosynthesis with placement of prosthetic materials

Exclusion Criteria:

* minor, can't or won't sign PIC, can't undergo surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: trimalleolar farcture lower extremity, requiring osteosynthesis and external fixation undergoing revision to internal fixation; osteosynthesis of upper extremity undergoing revision to receive inverse shoulder prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection | 3 months
  infection of osteosynthesis materials within 3 months after index procedure

SECONDARY OUTCOMES:
AE all grades, infections and all cause mortality during total follow up | 36 months
  AE all grades, infections and all cause mortality during total follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Helios Cuxhaven, Cuxhaven, Germany

IPD SHARING:
Plan to Share IPD: No